CLINICAL TRIAL: NCT05956743
Title: The Effect of Progressive Relaxation Exercise on Sleep Quality in Patients With Type 2 Diabetes
Brief Title: Progressive Relaxation Exercise on Sleep Quality in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ecem BİRER, NURSE, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MersinU-SBF-EB-01
Record Dates: First submitted 2023-07-14; First posted 2023-07-21 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: sleep quality; exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Initiation and Maintenance Disorders; Motor Activity | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: The research is carried out in two groups as control and intervention groups.
Masking Description: Participants and the researcher cannot be blinded due to the nature of the research. According to the randomized controlled research design, in this study, the groups of patients who would or would not be treated according to the simple random sampling method were determined.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): Intervention Group: A total of 6 weeks of planning will be made with the working group.
  1 week : Patients included in the study group and meeting the research criteria will be informed about the research. Pre-test data forms for each patient who accepted to participate in the study, Patient Identification Form, Pittsburgh Sleep Quality Index (PUKI) within 30 minutes will be collected.
  2.,3.,4.,5. week: Patients will practice a total of 12 progressive relaxation exercise sessions for 30 minutes, 3 times a week (Monday, Wednesday, Friday) for 4 weeks, accompanied by the training booklet and music player.
  6 week: In the last week of the application, individuals will be called to the hospital and in the Diabetes Polyclinic training room.A final test will be made by the researcher. The Pittsburgh Sleep Quality Index (PUKI) will be reapplied.
  Interventions: Other: progressive relaxation exercise sessions
- Sham group (Sham Comparator): 1 week: After informing Sham group patients about the research at the first interview, Patient Information Form, Pittsburgh Sleep Quality Index (PUKI) will be applied.
  In the 6th week of the study, individuals will be called to the hospital and the post-test Pittsburgh Sleep Quality Index (PUKI) will be re-administered by the researcher in the diabetes polyclinic training room.
  6 week: Since the study was terminated after the 6th week, a booklet and music player will be given to the patients. In addition, progressive relaxation exercise training will be given to the patients and the importance of using it in their lives will be explained.
  Interventions: Other: Sham

INTERVENTIONS:
Other: progressive relaxation exercise sessions — Intervention Group: A total of 6 weeks of planning will be made with the working group.
  1. week: Patients included in the study group and meeting the research criteria will be informed about the research. Pre-test data forms for each patient who accepted to participate in the study, Patient Identification Form, Pittsburgh Sleep Quality Index (PUKI) within 30 minutes will be collected.
  2. ,3.,4.,5. week: Patients will practice a total of 12 progressive relaxation exercise sessions for 30 minutes, 3 times a week (Monday, Wednesday, Friday) for 4 weeks, accompanied by the training booklet and music player.
  6. week: In the last week of the application, individuals will be called to the hospital and in the Diabetes Polyclinic training room. A final test will be made by the researcher. The Pittsburgh Sleep Quality Index (PUKI) will be reapplied.
  Arms: intervention group
Other: Sham — 1. week: After informing Sham group patients about the research at the first interview, Patient Information Form, Pittsburgh Sleep Quality Index (PUKI) will be applied.
  6. week: In the 6th week of the study, individuals will be called to the hospital and the post-test Pittsburgh Sleep Quality Index (PUKI) will be re-administered by the researcher in the diabetes outpatient training room. Since the study was terminated after the 6th week, a booklet and music player will be given to the patients. In addition, progressive relaxation exercise training will be given to the patients and the importance of using it in their lives will be explained.
  Arms: Sham group

SUMMARY:
The purpose of this study is to evaluate the effect of progressive relief exercise on sleep quality in patients with type 2 diabetes. Diabetes is among the diseases known as non-communicable or chronic diseases that occur as a result of the pancreas not producing enough insulin or the body's inability to use the insulin it produces and increasing the costs of care all over the world. Counseling and health education are among the key components of diabetes management. Diabetes management consists of drug therapy, self-management, medical nutrition therapy, exercise and education parameters, and sleep disorders are ignored in diabetes management. The slightest disruption to sleep patterns has definite and direct effects on daily life and general health. Therefore; stay healthy; Sleep is necessary renew and repair systems such as to renew and muscle systems. Inadequate sleep quality can lead to impaired cognition, and sleep quality is an important aspect of life. Sleep disturbance or poor sleep quality is higher in individuals with chronic disease. Sleep disturbance in diabetes is associated with higher HbA1c levels and diseases such as diabetes reduce sleep quality and regularity; It is known to cause sleep disorders. Especially in Type 2 Diabetes cases, sleep problems are common. Having a chronic illness like Type 2 Diabetes can have an impact on sleep quality and rate alone. Complementary and integrated applications such as progressive relaxation exercise, which is one of the cognitive behavioral techniques, have been frequently used in researches in the field of nursing, due to its effects such as relatively relieving tension and anxiety in skeletal muscles, facilitating the transition to sleep and helping to reduce sleep problems. Despite the differences in progressive muscle relaxation methods, studies have shown that progressive muscle relaxation has important results in improving sleep quality in individuals with chronic diseases. In this respect, it is predicted that progressive relaxation exercise may give positive results on sleep quality in individuals with diabetes.

DETAILED DESCRIPTION:
Diabetes is among the diseases known as non-communicable or chronic diseases that occur as a result of the pancreas not producing enough insulin or the body's inability to use the insulin it produces and increasing the costs of care all over the world. Worldwide, 537 million adults live with diabetes, and Type 2 Diabetes is the most common type of diabetes worldwide, accounting for approximately 90% of all diabetes cases. According to the Diabetes Epidemiological Study in Turkey data (TURDEP-I and II), the prevalence of diabetes increased from 7.2% to 13.7%. While there is a globally agreed target to halt the increase in diabetes by 2025, both the number of cases and the prevalence of diabetes continue to rise steadily over the past few decades. It is estimated that the total number of individuals with diabetes will increase to 643 million by 2030 and to 784 million by 2045. Counseling and health education are among the key components of diabetes management. Diabetes management consists of drug therapy, self-management, medical nutrition therapy, exercise and education parameters, and sleep disorders are ignored in diabetes management. diabetes association recently included sleep as a behavior to watch among adults living with diabetes in its 2019 and 2020 standards of care. Sleep; It is a periodic process in which physical activities are at the lowest level and the level of consciousness shows reversible changes. Sleep quality, which is one of the most important aspects of sleep; It is a complex phenomenon that is difficult to define and measure objectively. Sleep quality; It includes quantitative aspects of sleep such as sleep latency, duration of sleep, and the number of awakenings per night, and more subjective aspects such as sleep depth and restfulness. Sleep; It includes a multidimensional regeneration process, including physiological, psychological and social. For this reason, it is affected by positive/negative changes in the dimensions it covers. The slightest disruption to sleep patterns has definite and direct effects on daily life and general health. Therefore; stay healthy; Sleep is necessary to renew and repair systems such as neurological and muscle systems. Inadequate sleep quality can lead to impaired cognition, and sleep quality is an important aspect of life. Sleep disturbance or poor sleep quality is higher in individuals with chronic disease. Sleep disturbance in diabetes is associated with higher HbA1c levels and chronic diseases such as diabetes reduce sleep quality and regularity; It is known to cause sleep disorders. Individuals with uncontrolled diabetes often wake up sweating at night or due to nocturia. Controlling blood sugar with dietary changes, exercise, and medications can reduce sleep problems. Night movements or pain caused by the presence of neuropathy in the patient may also negatively affect sleep quality.Especially in Type 2 Diabetes cases, sleep problems are common. Having a chronic illness like Type 2 Diabetes can have an impact on sleep quality and rate alone. Sleep deprivation is a risk factor for impaired glucose tolerance, patients with diabetes have low sleep quality, there is a significant relationship between diabetes and sleep quality, and people with Type 2 Diabetes have poor sleep quality. Studies have determined that the probability of developing impaired fasting blood glucose in individuals is 6 times higher than in individuals who sleep an average of 6-8 hours at night and have good sleep quality. According to the report of the "American Academy of Sleep Medicine" center, the development or worsening of diabetes with sleep deprivation and sleep disorder there is a link between them. There are metabolic syndrome components such as hyperinsulinemia, central obesity, glucose intolerance in "Obstructive Sleep Apnea" which is a kind of sleep disorder. It is stated in the publications that "Obstructive Sleep Apnea" causes the development of diabetes by disrupting the glucose metabolism. Obstructive sleep apnea, short sleep duration, shift work, and insomnia are all associated with a higher risk of type 2 diabetes and may have worse outcomes for those with existing diabetes. Complementary and integrated applications such as progressive relaxation exercise, which is one of the cognitive behavioral techniques, have been frequently used in research in the field of nursing, due to its effects such as relatively relieving tension and anxiety in skeletal muscles, facilitating the transition to sleep and helping to reduce sleep problems.

Progressive relaxation is a method that provides relaxation throughout the body by regular voluntary and successive contraction and relaxation of large muscle groups in the human body. Purpose of progressive relaxation exercises; It is based on feeling the difference between tension and looseness in the body and learning to relax in our daily life. This method, which is applied in the form of stretching and relaxing the muscles, allows the patients to learn where their muscles are, what they are in the moment of tension, and the difference when the tension disappears. Benefits of progressive muscle relaxation in diabetes; It improves metabolic control, lowers blood sugar, lowers catecholamines and autonomic nerve activity. After relaxation, the patient will feel relaxed and relaxed, progressive relaxation body; will be able to make the mind calm and relaxed. Relaxation improves blood circulation, increases the secretion of endorphins and decreases the secretion of adrenal hormones, reduces stress and anxiety after the emergence of a positive attitude due to increased brain function, and facilitates sleep. Progressive relaxation exercises are a skill that can be taught by nurses and learned in both inpatient and outpatient settings that include the nurse's role as educator, caregiver, role model and patient advocate, and is included in the Classification of Nursing Interventions (NIC). Nurses' use of high-level nursing practices, such as training patients with relaxation exercises, improves the patient's self-management skills and provides symptom control. Despite the differences in progressive muscle relaxation methods, studies have shown that progressive muscle relaxation has important results in improving sleep quality in individuals with chronic diseases. In this respect, it is predicted that progressive relaxation exercise may give positive results on sleep quality in individuals with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes for at least 6 months
* Not having any disease causing insomnia and not using sleeping pills
* Willing to participate in the research
* 18 years and older
* Fluent in Turkish, Literate
* Understanding the given information and practicing the progressive relaxation exercise
* Related to vision, speech and hearing, which can interfere with the application of without disease,
* Not having a psychiatric diagnosis and not taking any medication for anxiety or depression
* Patients who have a music player or a personal mobile phone at home will be included in order to practice progressive relaxation exercises.

Exclusion Criteria:

* Those who do not agree to participate in the research
* Having any disease that causes insomnia and using sleeping pills
* Visual, speech and hearing impairments that can prevent the understanding of the given information and the implementation of the progressive relaxation exercise.

sick

* Having a psychiatric diagnosis and taking medication for anxiety or depression
* Do not have a music player or a personal mobile phone at home in order to practice progressive relaxation exercises.
* Patients working in shifts will not be included.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Four week
  The Pittsburgh Sleep Quality Index (PUKI) was developed(1989). The scale consists of 24 questions in total. 19 of these questions are answered by the individual and 5 of them are answered by the relative/roommate of the individual. Of these 5 questions and self-assessment questions, the last question, Question 19 (regarding the availability of a roommate or spouse), is used for clinical information only and is not included in the scoring. PUKI; The questions answered directly by the individual consist of 7 sub-components in which sleep duration, subjective sleep quality, sleep efficiency, sleep delay, degree of sleep disturbance in daytime work, and use of sleeping pills are evaluated. Each component is evaluated with a score between 0-3 and a total of 0-21 points can be obtained from the scale. An increase in the PUKI score means that the quality of sleep worsens. A total PUKI score of 5 or more is considered poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Diğdem LAFCI, Assoc. Dr., Principal Investigator — Mersin University
Locations (1):
- Nigde Training and Research Hospital, Niğde, Merkez/ Ni̇ğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No